CLINICAL TRIAL: NCT05926609
Title: A Placebo-Controlled, Single-Blind Sequential Study to Evaluate the Efficacy of EB-PA on Muscle Mass and Strength in Occasional Gym Goer
Brief Title: A Study to Evaluate the Efficacy of EB-PA on Muscle Mass and Strength in Occasional Gym Goers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: EB/230201/EB-PA/MMS
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Muscle Mass and Strength

STUDY DESIGN:
Intervention Model Description: Single-blind, placebo - controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EB-PA (Active Comparator): One capsule to be taken after breakfast once a day for 30 days
  Interventions: Dietary Supplement: EB-PA
- Placebo (Placebo Comparator): One capsule to be taken after breakfast once a day for 30 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EB-PA — 1 capsule to be taken after breakfast once a day
  Arms: EB-PA
Dietary Supplement: Placebo — 1 capsule to be taken after breakfast once a day
  Arms: Placebo

SUMMARY:
The present study is a placebo- controlled, single-blind sequential study. Total of 40 males aged between ≥ 18 years and ≤35 years will be screened. Assuming screen failure and dropout rate in this study, a minimum of 30 participants should complete the study. The treatment duration for all the study participants will be 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥18 to ≤ 35 years with moderate physical activity levels as per International Physical Activity Questionnaire (IPAQ-SF).
* Occasionally gym goer with a history of at least 1 month of training but not participating in the resistance-type activity for ≥3 months.
* Habitual non-veg eater
* Body mass index (BMI) 22 - 29.9 kg/ m2
* Waist Circumference 94-102 cm
* Ready to refrain from caffeinated products and intense strength/ endurance exercise for 24 hrs before the exercise lab visit.
* Fasting blood Glucose ≤ 125 mg/ dl
* Systolic Blood Pressure ≤ 129 mm Hg and Diastolic Blood Pressure ≤ 89 mm Hg
* TSH (thyroid stimulating hormone) ≥0.4 and ≤ 4.9 mIU/L

Exclusion Criteria:

* Engaged in structured weight training for more than 12 months before screening.
* Presence of chronic disease
* Changes in body weight of more than 4.5 kg (10 pounds) in the past three months
* Individuals with uncontrolled hypertension
* Known cases of Type II Diabetes mellitus
* History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic, or neurologic disorders
* Individuals who have any other disease or condition or are using any medication that, in the investigator's judgment would put them at unacceptable risk for participation in the study or may interfere with evaluations or non-compliance with treatment or visits
* Individuals who have been part of a clinical trial within 90 days before the screening
* Individuals who have used whey or other supplements anytime in the last 3 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) from baseline on | Day 31
  Improvement in muscle strength as assessed by isokinetic peak torque (measured during knee extension and flexion)
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) from baseline on | Day 61
  Improvement in muscle strength as assessed by isokinetic peak torque (measured during knee extension and flexion)

SECONDARY OUTCOMES:
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Increase in the lower-body strength (Peak anaerobic power output (PAPw)) as assessed by a vertical jump test
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Improvement in upper body strength as assessed by medicine ball throw test
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  The flexibility of the hamstrings as assessed using the V sit-and-reach test
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Improvement in muscle mass as indicated by an increase in fat-free mass (FFM) by DXA
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Decrease in central obesity as indicated by a decrease in android fat percentage by DXA.
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Improvement in metabolic health as indicated by the waist-to-height ratio (WHtR)
To assess the effect of 30 days (Baseline to end of treatment period) administration of investigational product (IP) on | Day 0, Day 31 and Day 61
  Improves muscle protein synthesis as assessed by an increase in serum insulin at 0, 1 & 3 hours post IP administration.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Dr. Kumta Solanki's Clinic, Mumbai, Maharashtra
  - Dr. Preeti Bawaskar's Clinic, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided